CLINICAL TRIAL: NCT05232838
Title: US Pilot Study to Evaluate the Safety and Effectiveness of the CereVasc® eShunt® System in the Treatment of Normal Pressure Hydrocephalus
Brief Title: US Pilot Study of the CereVasc® eShunt® System in Normal Pressure Hydrocephalus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CereVasc Inc (Industry)
Collaborators: AlvaMed, Inc. (Industry); Simplified Clinical Data Systems, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0016
Record Dates: First submitted 2022-01-06; First posted 2022-02-10 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Hydrocephalus, Normal Pressure; Hydrocephalus
Keywords: eShunt; Minimally invasive shunt; Endovascular shunt
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Hydrocephalus

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Arm (Experimental): The Treatment Arm receives the eShunt Implant.
  Interventions: Device: eShunt Implant

INTERVENTIONS:
Device: eShunt Implant — The eShunt System is intended to shunt cerebrospinal fluid from the intracranial subarachnoid space to the venous system for the treatment of patients with normal pressure hydrocephalus, reducing disability due to symptoms including one or more of gait disturbance, cognitive dysfunction and urinary incontinence.

SUMMARY:
The eShunt® System is a minimally invasive method of treating communicating hydrocephalus. The eShunt System includes a proprietary eShunt Delivery System and the eShunt Implant, a permanent implant deployed in a minimally invasive, neuro-interventional procedure. The eShunt System is intended to shunt cerebrospinal fluid from the intracranial subarachnoid space to the venous system for the treatment of patients with normal pressure hydrocephalus, reducing disability due to symptoms including one or more of gait disturbance, cognitive dysfunction and urinary incontinence.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, open-label, multi-center, pilot study in subjects with normal pressure hydrocephalus for whom a traditional cerebrospinal fluid (CSF) shunt implant is indicated.

Up to 50 subjects will receive the eShunt Implant at up to 12 investigational sites. It is anticipated that up to 250 patients may need to be enrolled (consented) in order to result in 50 subjects who qualify according to the inclusion/exclusion criteria. Subjects will return for five follow-up visits in the first year and then continue to attend visits every six months until the study is closed or up to five years post-implantation.

The study objectives are to demonstrate safety of the eShunt Procedure, as well as demonstrate safety and efficacy of the eShunt Implant in a small sample of patients. Subjects will be followed long-term; primary analysis results will be used to support additional studies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 65-85 years old for whom traditional CSF shunt placement is indicated based upon a diagnostic normal pressure hydrocephalus (NPH) evaluation
2. Patient or legally authorized representative is able and willing to provide written informed consent
3. History or evidence of gait impairment duration ≥6 months
4. Clinical presentation consistent with NPH including 2 or more of the clinical triad (i.e., history of gait disturbance, progressive mental deterioration, and urinary urgency or incontinence), together with:

   1. Brain MRI signs of ventricular enlargement disproportionate to cerebral atrophy (Evans' Index >0.3) and the absence of severe hippocampal atrophy
   2. Pre-procedure spinal tap test or lumbar drain with subsequent gait disturbance improvement (Timed Up and Go Test) of at least 20%
   3. CSF opening pressure ≥8 cmH2O
   4. Baseline cognitive evaluation assessed by Montreal Cognitive Assessment (MoCA) test score ≥12
5. Pre-procedure MRI confirmation of anatomy suitable for eShunt Procedure, as described in Section 1.8.3.4.2 and confirmed by subject screening committee (SSC)
6. Pre-procedure CT confirmation of anatomy suitable for eShunt Procedure, as described in Section 1.8.3.4.2 and confirmed by SSC

Exclusion Criteria:

1. Unable to walk 10 meters (33 feet) with or without an assistive device
2. Signs or symptoms of obstructive hydrocephalus
3. Active systemic infection or infection detected in CSF
4. Prior or existing shunts, endoscopic third ventriculostomy, or any previous surgical intervention for hydrocephalus
5. Hypersensitivity or contraindication to heparin or radiographic contrast agents which cannot be adequately pre-medicated, desensitized or where no alternative is available
6. Occlusion or stenosis of the internal jugular vein
7. Venous distension in the neck on physical exam
8. Atrial septal defect or patent foramen ovale identified on cardiac echocardiogram
9. History of bleeding diatheses, coagulopathy or will refuse blood transfusion in cases of emergency
10. Stroke or transient ischemic attack within 180 days of eShunt Procedure
11. Presence of a deep vein thrombosis superior to the popliteal vein
12. International Normalized Ratio (INR) or Partial Thromboplastin Time (PTT) results outside of normal range (INR 0.8-1.4; PTT 25-35 seconds)
13. Presence of a posterior fossa tumor or mass
14. Life expectancy < 1 year
15. Currently participating in another investigational drug or device trial that could conflict with study data collection or follow-up
16. Other medical illnesses that may cause the patient to be non-compliant with the protocol or confound data interpretation
17. Unwilling or unable to comply with follow-up requirements

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Device and/or procedure-related serious adverse events (SAEs) | 90 days following eShunt Implant deployment
  Rate of occurrence of device and/or procedure-related serious adverse events (SAEs)

SECONDARY OUTCOMES:
Number of participants with abnormal MRI findings | 90 days following eShunt Implant deployment
  Number of participants with abnormal MRI findings and descriptive summaries of findings
Number of participants with abnormal CT findings | 90 days following eShunt Implant deployment
  Number of participants with abnormal CT findings and descriptive summaries of findings
Number of participants with clinically significant abnormal complete blood count (CBC) results | 90, 180, and 365 days following eShunt Implant deployment
  Number of participants with clinically significant abnormal results and descriptive summaries of CBC results
Number of participants with clinically significant abnormal blood chemistry results | 90, 180, and 365 days following eShunt Implant deployment
  Number of participants with clinically significant abnormal findings and descriptive summaries of blood chemistry results
Number of participants with clinically significant abnormal neurological exam findings | 90, 180, and 365 days following eShunt Implant deployment and at study completion
  Number of participants with clinically significant abnormal findings and descriptive summaries of neurological exam findings
Number of participants with adverse events | 90, 180 and 365 days following eShunt Implant deployment and at study completion
  Tabulation of all adverse events
Change in gait compared to baseline | 90, 180 and 365 days following eShunt Implant deployment
  Change in gait compared to baseline as measured by the duration in seconds of the Timed Up and Go Test (shorter durations indicate improvement (increased mobility))
Change in cognitive ability compared to baseline | 90, 180 and 365 days following eShunt Implant deployment
  Change in cognitive ability compared to baseline as measured by Montreal Cognitive Assessment (MoCA) scores (scores range from 0-30; higher scores indicate improvement (less cognitive disability))
Change in urinary symptoms compared to baseline | 90, 180 and 365 days following eShunt Implant deployment
  Change in urinary symptoms compared to baseline as measured by the Neurogenic Bladder Symptom Score (NBSS) (scores range from 0-28; lower scores indicate improvement (fewer symptoms))
Change in Modified Rankin Scale compared to baseline | 90, 180 and 365 days following eShunt Implant deployment
  Change in degree of disability compared to baseline as measured by Modified Rankin Scale (mRS) scores (scores range from 0-6; lower scores indicate improvement (less disability))

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Yale University, New Haven, Connecticut
  - Baptist Health, Jacksonville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Research Foundation, Lexington, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University at Buffalo,, Buffalo, New York
  - NYU Langone Health, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Rhode Island Hospital, Providence, Rhode Island
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heilman CB, Basil GW, Beneduce BM, Malek AM. Anatomical characterization of the inferior petrosal sinus and adjacent cerebellopontine angle cistern for development of an endovascular transdural cerebrospinal fluid shunt. J Neurointerv Surg. 2019 Jun;11(6):598-602. doi: 10.1136/neurintsurg-2018-014445. Epub 2019 Jan 9. PMID 30626626
- [Background] Lylyk P, Lylyk I, Bleise C, Scrivano E, Lylyk PN, Beneduce B, Heilman CB, Malek AM. First-in-human endovascular treatment of hydrocephalus with a miniature biomimetic transdural shunt. J Neurointerv Surg. 2022 May;14(5):495-9. doi: 10.1136/neurintsurg-2021-018136. Epub 2021 Dec 3. PMID 34862267
- [Background] Welk B, Morrow S, Madarasz W, Baverstock R, Macnab J, Sequeira K. The validity and reliability of the neurogenic bladder symptom score. J Urol. 2014 Aug;192(2):452-7. doi: 10.1016/j.juro.2014.01.027. Epub 2014 Feb 8. PMID 24518764
- [Background] Welk B, Lenherr S, Elliott S, Stoffel J, Gomes CM, de Bessa J, Cintra LKL, Myers JB; Neurogenic Bladder Research Group. The creation and validation of a short form of the Neurogenic Bladder Symptom Score. Neurourol Urodyn. 2020 Apr;39(4):1162-1169. doi: 10.1002/nau.24336. Epub 2020 Mar 20. PMID 32196732
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Derived] Amllay A, Matouk CC. A Paradigm Shift in Hydrocephalus Management: The Promise of Endovascular Cerebrospinal Fluid Diversion. Cardiol Rev. 2025 Jul-Aug 01;33(4):294-297. doi: 10.1097/CRD.0000000000000886. Epub 2025 Mar 26. PMID 40135887